CLINICAL TRIAL: NCT06298942
Title: Naturally Banded Versus Synthetic Banding of Sleeve Gastrectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Alaa Mstafa Hassan Sewefy, professor & consultant of general surgery,, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fac.med.24.9
Record Dates: First submitted 2024-02-21; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Obesity, Morbid
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- natural band (Experimental): to use an round ligament as a natural band in stead of synesthetic band with sleeve gastrectomy
  Interventions: Procedure: natural band
- silicone band (Active Comparator): to use a synesthetic band with sleeve gastrectomy
  Interventions: Procedure: silicone band

INTERVENTIONS:
Procedure: natural band — to use the round ligament as a natural band in stead of synesthetic band with sleeve gastrectomy
  Arms: natural band
Procedure: silicone band — to use synesthetic band with sleeve gastrectomy
  Arms: silicone band

SUMMARY:
to compare banding sleeve gastrectomy using silicone ring Versus using natural flap ( round ligament of the liver)

DETAILED DESCRIPTION:
to compare banding sleeve gastrectomy using silicone ring Versus using natural flap ( round ligament of the liver) as regard weight loss, complications rat and cost

ELIGIBILITY:
Inclusion Criteria:

* obese patients with BMI more than 40 with or without co-morbidity or more than 35 with co-morbidity
* patients fit for laparoscopic surgery
* give approval to share in the study

Exclusion Criteria:

* patients refused to share in the study
* patients unfit for surgery
* patients aged less than 18 and older than 65
* patient with previous upper abdominal surgery either for obesity or other diseases
* revisional bariatric procedures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-03-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
total cost | 12 hours
  total operative cost in Egyptian pound (LE)
food intolerance | 1 year
  food intolerance at one year food tolerance arabic score questionnaire

SECONDARY OUTCOMES:
%EWL | 1 year
  percentage of weight loss at one year measured as (initial weight - follow-up weight) / (initial weight - bodyweight at a BMI of 25 kg/ m2) x 100
complications rate | 1 year
  the incidence of early and late complications according to Clavien-Dindo (CD)
improvement of comorbidities | 1 year
  the incidence of improvement of comorbidities